CLINICAL TRIAL: NCT00701623
Title: Clinical Efficacy of Product Alimax ® (Sodic Heparin) in Treatment of Burns: Comparative Study of Raw Materials Between Two Suppliers
Brief Title: Sodic Heparin Effectiveness of the Treatment of Burns
Acronym: Heparin
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Azidus Brasil (Industry)
Responsible Party: Principal Investigator, Azidus Brasil, Principal Investigator Dr. Alexandre Frederico, Azidus Brasil
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HEPCRI0208
Record Dates: First submitted 2008-06-17; First posted 2008-06-19 (Estimated); Last update posted 2022-11-03 (Actual); Status verified 2022-11

CONDITIONS: Burns
Keywords: sodium heparin; burns of the skin
MeSH Terms: conditions — Burns | interventions — Heparin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): patients treated with heparin
  Interventions: Drug: heparin
- 2 (Experimental): Patients treated with heparin
  Interventions: Drug: heparin
- 3 (Active Comparator): patients treated with folder water directly on the injured area
  Interventions: Drug: folder water

INTERVENTIONS:
Drug: heparin — patients will receive the application of one of two types of heparin directly on the injured area
  Arms: 1
Drug: heparin — patients will receive the application of one of two types of heparin directly on the injured area
  Arms: 2
Drug: folder water — patients will receive the application of folder water directly on the injured area
  Arms: 3

SUMMARY:
Burns are injuries caused by agents thermal, chemical, electrical or radioactive who act in the tissue lining of the human body and may partially or totally destroy the skin and its annexes, to the deeper layers, as subcutaneous tissue, muscles, tendons and bones .

Studies show that topical heparin has, in addition to the already known anticoagulant activity, anti-inflammatory properties, analgesic, and neoangiogenic, stimulating blood flow and increasing the repair of the fabric as well as the restoration of collagen and reepiteliztion. Moreover, the use of heparin reduces the need for painful medical procedures, as debridations, surgeries and transplants The intention of this work is to verify the effectiveness and safety of sodium heparin in the treatment of burns of the skin.

DETAILED DESCRIPTION:
Patients with burns that come to the emergency room will be informed about the

Inclusion Criteria

* Patients aged above 12 years who have suffered thermal burns of 2nd degree burns or mixed 2 and 3 degrees in up to 10% of body surface and indication of outpatient treatment.

Exclusion Criteria

* Area burned more than 10% of body surface
* the presence of the 3 rd degree burns
* burns in the face or genitals
* burns in poly-traumatized
* respiratory injury
* disorders of coagulation
* thrombocytopenia
* erosive gastro cases
* clinically relevant bleeding
* hypersensitivity to anticoagulants
* liver disease
* nephropathy
* diabetes
* 35
* serious allergy
* descontrole emotional
* pregnancy
* anemia

ELIGIBILITY:
Inclusion Criteria:

* Patients aged above 12 years who have suffered thermal burns of 2nd degree burns or mixed 2 and 3 degrees in up to 10% of body surface and indication of outpatient treatment.

Exclusion Criteria:

* Area burned more than 10% of body surface
* the presence of the 3 rd degree burns
* burns in the face or genitals
* burns in poly-traumatized
* respiratory injury
* disorders of coagulation
* thrombocytopenia
* erosive gastro cases
* clinically relevant bleeding
* hypersensitivity to anticoagulants
* liver disease
* nephropathy
* diabetes
* 35
* serious allergy
* descontrole emotional
* pregnancy
* anemia

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-06 (Actual); Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Primary: immediate decrease in pain. Secondary: analgesic request for 10 minutes after application of heparin, signs of intolerance and adverse events. | healing

CONTACTS AND LOCATIONS:
Locations (1):
- LAL Clinica PPesquisa e Desenvolvimento, Valinhos, São Paulo, Brazil